CLINICAL TRIAL: NCT03995953
Title: Developing and Testing a Multi-level Package of Interventions for an Integrated Care Delivery Model of HIV Prevention and Treatment Targeting Adolescent Girls in Zambia
Brief Title: Integrated Care Delivery of HIV Prevention and Treatment in AGYW in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Population Council (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1UG3HD096908-01 (NIH); 1UG3HD096908-01 (NIH)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: HIV prevention; HIV treatment; Zambia
MeSH Terms: interventions — Palliative Care; Ambulatory Care Facilities

STUDY DESIGN:
Intervention Model Description: Based on their residence in the catchment areas of the six selected study clinics, AGYW participants, stratified by age group and HIV status, will be randomized into the following three treatment arms: no intervention, the SHIELD intervention, and the SHIELD intervention and IWC clinics. The sample size was calculated assuming conventional specifications (power = .80, alpha = .05, two-sided tests) and based on the primary endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 2 control clinics, and their associated catchment areas, with no intervention at the clinic or community level
- SHIELD: Community-based behavioral intervention (Experimental): 2 clinics, and their associated catchment areas, where participants attend modules designed to educate and empower adolescent girls and young women (AGYWs) and their caregivers, along with attendance at community-based youth clubs to foster peer support.
  Interventions: Behavioral: SHIELD intervention (Support for HIV Integrated Education, Linkages to care, and Destigmatization)
- SHIELD: Community- based behavioral intervention & IWC Clinic (Experimental): 2 clinics, and their associated catchment areas, where participants and their caregivers receive the Support for HIV Integrated Education, Linkages to care, and Destigmatization (SHIELD) intervention along with the coupled benefits of having an integrated wellness care (IWC) clinic within health facilities where adolescent girls and young women (AGYWs) can receive sexual and reproductive health services, including HIV testing and treatment, family planning, sexually transmitted disease screening and treatment, and human papilloma virus (HPV) vaccination.
  Interventions: Behavioral: SHIELD intervention (Support for HIV Integrated Education, Linkages to care, and Destigmatization); Other: Integrated wellness care (IWC) clinics

INTERVENTIONS:
Behavioral: SHIELD intervention (Support for HIV Integrated Education, Linkages to care, and Destigmatization) — The SHIELD intervention includes a three-session, six-module program for AGYW that increases knowledge, skills, and self-efficacy to engage along the HIV prevention and care continuum, and a two-session, four-module program for caregivers to increase social support. In addition, the SHIELD intervention includes youth clubs to foster peer support.
  Arms: SHIELD: Community- based behavioral intervention & IWC Clinic; SHIELD: Community-based behavioral intervention
Other: Integrated wellness care (IWC) clinics — IWC clinics will be created within health facilities where AGYWs can receive sexual and reproductive health services, including HIV testing and treatment, family planning, sexually transmitted disease screening and treatment, and HPV vaccination in a youth-friendly environment.
  Arms: SHIELD: Community- based behavioral intervention & IWC Clinic

SUMMARY:
The study team will test a multilevel package of interventions to connect adolescent girls and young women (AGYW) with a source of regular care to provide a sustainable platform for successful implementation of regular human immunodeficiency virus (HIV) testing and support for linkage to care, retention in care, and adherence to antiviral treatment. Interventions will include integrated wellness care (IWC) clinics and the SHIELD intervention (Support for HIV Integrated Education, Linkages to care, and Destigmatization) to educate and empower AGYW and their families, and to create community-based youth clubs to foster peer support. A cluster randomized controlled trial will be implemented where AGYW participants, stratified by age group and HIV status, will be randomized based on their residence within the six study clinic catchment areas, into the following intervention arms: no intervention, the SHIELD intervention, and the SHIELD intervention and IWC clinics.

DETAILED DESCRIPTION:
The SHIELD intervention aims to improve HIV prevention and care for adolescent girls and young women (AGYW) in Zambia. It is based on social cognitive theory and includes a program for AGYW to increase knowledge, skills, and self-efficacy, as well as a program for family members to increase social support. The intervention also incorporates youth clubs facilitated by peer navigators and integrated wellness clinics (IWC) for sexual and reproductive health services. It will be tailored for five distinct groups based on age and HIV status, with modules covering HIV prevention and treatment, wellness, sexual health, stigma reduction, and healthcare access.

IWC clinics will be established in existing government health facilities, following a model similar to cervical cancer screening clinics. Standard operating procedures (SOPs) will be developed for HIV, HPV vaccination, and sexual and reproductive health services.

Time and motion methodology will monitor AGYW clinic visits to identify areas for improvement. To establish a sampling frame, the study team will identify six clinics in Lusaka, map neighborhoods within the selected clinic catchment areas, and recruit AGYW through household visits by peer navigators.

The HIV-/u cohort will include females aged 10-20 years with self-reported HIV-negative or unknown status. They must not be pregnant or planning pregnancy, be willing to sign a medical records release, plan to reside in the area for 18 months, and not be part of other formative research activities. The study will recruit 1,000 HIV-/u AGYW, with equal numbers in age ranges 10-12, 13-15, and 16-20.

The HIV+ cohort will consist of females aged 16-24 years, diagnosed with HIV within the past 3 years, and meeting the same additional criteria as the HIV-/u cohort. The study will enroll 800 HIV+ AGYW, with equal representation among 16-20 and 21-24 age groups.

AGYW will be encouraged to select caregivers who will participate in some of the education sessions. The role of the caregiver is to support AGYW. Primary and secondary outcomes will be reported for AGYW only.

Data collection will use electronic tablets with pre-loaded software and instruments in multiple languages. Voice-enabled components and self-administration options will be available for sensitive questions. Instruments will be pretested with AGYW and caregivers. The study team will abstract data from clinic records with support from the Zambian Ministry of Health, conducting pilot data abstraction and staff training to ensure high-quality data for the study.

Key aspects of the intervention include tailored education modules for AGYW and caregivers, youth clubs led by peer navigators, and integrated wellness clinics offering comprehensive sexual and reproductive health services.

The SHIELD study aims to improve HIV prevention and care for AGYW in Zambia by addressing knowledge, skills, self-efficacy, social support, and healthcare access through a comprehensive, theory-based intervention. By combining education, social support, and improved healthcare services, the researchers hope to make significant strides in reducing HIV transmission and improving health outcomes for adolescent girls and young women in Zambia.

ELIGIBILITY:
Inclusion Criteria:

HIV negative or unknown cohort

* Female
* 10 to 20 years of age
* self-report HIV status as negative or unknown (no HIV testing within the past 6 months
* not pregnant, does not suspect pregnancy, and does not express a desire to become pregnant over the next 18 months
* is willing to sign a release for medical records (to obtain clinic data on service use)
* plans to reside in the current location for the next 18 months
* has not been part of the other planned formative research activities

HIV positive cohort

* Female
* 16 to 24 years of age
* diagnosed with HIV within the past 3 years or newly diagnosed at the time of the study
* not pregnant, does not suspect pregnancy, and does not express a desire to become pregnant over the next 18 months
* is willing to sign a release for medical records (to obtain clinic data on service use)
* plans to reside in the current location for the next 18 months
* has not been part of the other planned formative research activities

Exclusion Criteria:

* pregnant

Ages: 10 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2150 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujha Subramanian, PhD, Principal Investigator — Implenomics
Locations (1):
- Population Council, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the data will be placed in an NIH electronic database that could be used by researchers outside our study team who are interested in using it to answer questions about access to youth-friendly health services in Zambia. Responses will be inputted after they have been stripped of identifiers such as name, so that it may be used and shared for future research. This research will provide useful feedback for behavior of adolescents at risk or living with HIV in the United States.

REFERENCES:
- [Derived] Scanlon SL, Blackburn NA, Beizer J, Mulenga DM, Nyblade L, Roberts ST, Chelwa N, Mbizvo M, Subramanian S. Comparison of sexual risk behaviors among Zambian adolescent girls and young women living with and without HIV. Reprod Health. 2025 Sep 30;22(1):174. doi: 10.1186/s12978-025-02147-2. PMID 41029779
- [Derived] Blackburn NA, Scanlon SL, Beizer J, Chelwa N, Nyblade L, Roberts ST, Phiri L, Mulenga D, Mbizvo M, Subramanian S. The Implementation and Costs To Deliver a youth-friendly multi-component Program Addressing Stigma, HIV, and Linkage To Care for Adolescent Girls and Young Women in Lusaka, Zambia. AIDS Behav. 2025 Jul;29(7):2179-2188. doi: 10.1007/s10461-025-04682-2. Epub 2025 Mar 20. PMID 40111579
- [Derived] Subramanian S, Edwards P, Roberts ST, Musheke M, Mbizvo M. Integrated Care Delivery for HIV Prevention and Treatment in Adolescent Girls and Young Women in Zambia: Protocol for a Cluster-Randomized Controlled Trial. JMIR Res Protoc. 2019 Oct 3;8(10):e15314. doi: 10.2196/15314. PMID 31584004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited adolescent and young women (AGYWs) from 6 clinic sites in the Lusaka, Zambia area. AGYWs were the main participants in the clinical trial and caregivers were recruited in a support capacity for AGYWs.
Pre-assignment Details: Assigned to HIV+ or HIV-/u depending on their HIV status at the time of enrollment.
Groups:
- Control HIV+ AGYW: HIV+ AGYW allocated to the control arm
- Control HIV+ Caregiver: Caregivers selected by HIV+ AGYW in the control arm.
- Control HIV- AGYW: HIV- AGYW allocated to the control arm
- Control HIV- Caregivers: Caregivers selected by HIV- AGYW in the control arm.
- SHIELD HIV+ AGYW: HIV+ AGYW allocated to the SHIELD only arm.
- SHIELD HIV+ Caregivers: Caregivers selected by HIV+ AGYW in the SHILED only arm.
- SHEILD HIV- AGYW: HIV- AGYW allocated to the SHIELD only arm
- SHIELD HIV- Caregivers: Caregivers selected by HIV- AGYW allocated to the SHIELD only arm.
- SHIELD+IWC HIV+ AGYW: HIV+ AGYW allocated to the SHIELD + IWC arm
- SHIELD+IWC HIV+ Caregivers: Caregiver selected by HIV+ AGYW in the SHIELD+IWC arm.
- SHIELD+IWC HIV- AGYW: HIV- AGYW allocated to the SHIELD+IWC arm.
- SHIELD+IWC HIV- Caregivers: Caregivers selected by HIV- AGYW in the SHIELD+IWC arm.
Period: Overall Study
Arm/Group | Control HIV+ AGYW | Control HIV+ Caregiver | Control HIV- AGYW | Control HIV- Caregivers | SHIELD HIV+ AGYW | SHIELD HIV+ Caregivers | SHEILD HIV- AGYW | SHIELD HIV- Caregivers | SHIELD+IWC HIV+ AGYW | SHIELD+IWC HIV+ Caregivers | SHIELD+IWC HIV- AGYW | SHIELD+IWC HIV- Caregivers
Started | 177 | 154 | 198 | 194 | 171 | 150 | 201 | 197 | 175 | 139 | 201 | 193
6 Months | 137 | 88 | 177 | 125 | 139 | 92 | 181 | 149 | 148 | 83 | 179 | 136
12 Months | 153 | 100 | 175 | 162 | 147 | 106 | 184 | 166 | 145 | 103 | 178 | 152
Completed | 153 | 100 | 175 | 162 | 147 | 106 | 184 | 166 | 145 | 103 | 178 | 152
Not Completed | 24 | 54 | 23 | 32 | 24 | 44 | 17 | 31 | 30 | 36 | 23 | 41
Not completed — Death | 3 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 54 | 3 | 32 | 5 | 44 | 0 | 31 | 8 | 36 | 5 | 41
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 0
Not completed — Health Issues | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Relocated | 11 | 0 | 16 | 0 | 14 | 0 | 16 | 0 | 14 | 0 | 15 | 0

BASELINE CHARACTERISTICS:
Population: The clinical trial only enrolled two cohorts of adolescent girls and young women (AGYW) between the ages of 10 and 24 living in Zambia (HIV-/u and HIV+) as well as caregivers who were only meant to serve as support for AGYW during education sessions.
Groups:
- AGYW Control: One-time Education (AGYW)
- AGYW SHIELD Only: SHIELD Intervention (AGYW)
- AGYW SHIELD + IWC Clinic: SHIELD Intervention and Integrated Wellness Clinic (AGYW)
- Caregiver Control: Caregivers appointed by those in AGYW Control.
- Caregiver SHIELD Only: Caregivers appointed by those in AGYW SHIELD Intervention.
- Caregiver SHIELD + IWC Clinic: Caregivers appointed by those in AGYW SHIELD Intervention and Integrated Wellness Clinic.
- Total: Total of all reporting groups
Arm/Group | AGYW Control | AGYW SHIELD Only | AGYW SHIELD + IWC Clinic | Caregiver Control | Caregiver SHIELD Only | Caregiver SHIELD + IWC Clinic | Total
Number analyzed (Participants) | 375 | 372 | 376 | 348 | 347 | 332 | 2150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 219 | 197 | 194 | 0 | 0 | 0 | 610
  Between 18 and 65 years | 156 | 175 | 182 | 341 | 340 | 324 | 1518
  >=65 years | 0 | 0 | 0 | 7 | 7 | 8 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (3.8) | 18.1 (3.8) | 18.0 (3.8) | 37.3 (11.3) | 37.7 (11.8) | 36.6 (11.9) | 27.2 (12.8)
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Total number of participants to be divided out by HIV status
  years
    HIV+: number analyzed (Participants) | 177 | 171 | 175 | 154 | 150 | 139 | 966
    HIV+ | 20.8 (2.5) | 21.0 (2.5) | 21.0 (2.3) | 39.8 (11.7) | 39.2 (11.7) | 38.5 (12.2) | 29.3 (12.3)
    HIV-/U: number analyzed (Participants) | 198 | 201 | 201 | 194 | 197 | 193 | 1184
    HIV-/U | 15.3 (2.7) | 15.6 (2.9) | 15.5 (2.9) | 35.4 (10.7) | 36.6 (11.7) | 35.3 (11.4) | 25.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 375 | 372 | 376 | 326 | 324 | 314 | 2087
  Male | 0 | 0 | 0 | 22 | 23 | 18 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 375 | 372 | 376 | 348 | 347 | 332 | 2150
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 375 | 372 | 376 | 348 | 347 | 332 | 2150
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 375 | 372 | 376 | 348 | 347 | 332 | 2150
HIV Status [Count of Participants; unit: Participants]
  HIV+ | 177 | 171 | 175 | 154 | 150 | 139 | 966
  HIV-/u | 198 | 201 | 201 | 194 | 197 | 193 | 1184

OUTCOME MEASURES:

1. Primary Outcome: HIV Testing
Description: Proportion of cohort not living with HIV that self-reported being tested for HIV in the past 6 months.
Time Frame: 6 months
Population: Adolescent Girls and Young Women not living with HIV in Lusaka, Zambia. The 6-month data collection was impacted by the COVID-19 pandemic and restrictions that were in place. We were unable to contact all of the participants we had enrolled at baseline as a result of pandemic restrictions which also caused participants to move away from their original enrollment catchment area. The reduction in participants should not be interpreted as drop-outs or those lost to follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control Group
- SHIELD Only: SHIELD Education Sessions
- SHIELD + IWC Clinic: SHIELD Sessions and Integrated Wellness Clinic
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 177 | 181 | 179
Participants | 33 | 52 | 139

2. Primary Outcome: HIV-/u Proportion Tested for HIV in the Past 6 Months
Description: Proportion of cohort not living with HIV that self reported being tested for HIV in past 6 months.
Time Frame: 12 months
Population: Adolescent Girls and Young Women not living with HIV in Lusaka, Zambia. The 12-month data collection occurred after COVID-19 restrictions had been lifted. The participant count increases from the 6-month count because we were able to contact participants we had previously been unable to reach and participants had moved back to their original enrollment catchment area and could be included in the participant count.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 175 | 184 | 178
Participants | 40 | 95 | 125

3. Primary Outcome: Retention in Care
Description: HIV+ cohort proportion with at least one visit during the 12-months follow-up. Data were not collected from any participant due to COVID 19 pandemic and associated restrictions, and will not be collected in the future.
Time Frame: 12 months
Population: Data were not collected from any participant due to COVID 19 pandemic and associated restrictions, and will not be collected in the future.
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: HIV+ Proportion With Undetectable Viral Load at 12 Months
Description: Proportion of cohort living with HIV who had an undetectable (less than 40 copies/mL) viral load
Time Frame: At 12 months since study initiation
Population: Adolescent Girls and Young Women living with HIV in Lusaka, Zambia.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Control adolescent Girls and Young Women living with HIV in Lusaka, Zambia
- SHIELD Only: SHIELD education sessions among adolescent Girls and Young Women living with HIV in Lusaka, Zambia
- SHIELD + IWC: SHIELD sessions and Integrated Wellness Clinic among adolescent Girls and Young Women living with HIV in Lusaka, Zambia
Arm/Group | Control | SHIELD Only | SHIELD + IWC
Number analyzed (Participants) | 151 | 143 | 141
Participants | 99 | 74 | 76

5. Secondary Outcome: HIV Risk Behavior - Delay in First Intercourse
Description: Self-reported age of first intercourse among HIV-/u cohort.
Time Frame: Baseline
Population: Zambian Adolescent and Young Women not living with HIV. The reason why the Overall Number of Participants Analyzed is substantially smaller than other categories is because questions related to sexual behavior and activity can only be asked to individuals aged 15 and over in Zambia. Our HIV-/u cohort is the cohort that enrolled participants between the ages of 10 and 26 and would, therefore, be most affected by the age restrictions in place for sexual behavior questions.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 40 | 48 | 51
years | 16.48 (2.36) | 16.85 (1.70) | 16.88 (1.63)

6. Secondary Outcome: HIV Risk Behavior - Delay in First Intercourse
Description: Self reported age of first intercourse among HIV-/u cohort.
Time Frame: 6 months
Population: Zambian Adolescent and Young women not living with HIV. The reason for seeing inconsistent participant sums for "6 month" row is because a fewer number of participants were surveyed/tested because of COVID and individuals leaving the area.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Control: One-time education
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 49 | 56 | 56
years | 17.10 (1.73) | 16.95 (1.76) | 16.94 (1.66)

7. Secondary Outcome: HIV Risk Behavior - Delay in First Intercourse
Description: HIV-/u self reported age of first intercourse.
Time Frame: 12 months
Population: Self-reported age of first intercourse among HIV-/u cohort. Reported values reflect results for those aged 16 and older since asking questions related to sexual behavior to those aged 15 and below in Zambia is illegal.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 56 | 68 | 61
years | 17.22 (1.70) | 17.20 (2.04) | 17.28 (1.45)

8. Secondary Outcome: HIV Risk Behavior - Reduction in Sexual Partners
Description: Self reported number of casual partners in the last 3 months among HIV-/u cohort.
Time Frame: Baseline
Population: Zambian Adolescent and Young Women not living with HIV. Questions related to sexual behavior and activity cannot be asked to individuals aged 15 and under in Zambia. Our HIV-/u cohort enrolled participants between the ages of 10 and 24 and would, therefore, be most affected by the age restrictions in place for sexual behavior questions. The number reported reflects the mean number of casual partners for all respondents who reported at least 1 sexual partner in each intervention group.
Measure: Mean (Full Range); unit: Mean of Casual Partners
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 39 | 48 | 50
Mean of Casual Partners | 1.14 [0 to 4] | 1.10 [0 to 4] | 1.06 [0 to 4]

9. Secondary Outcome: HIV Risk Behavior - Reduction in Sexual Partners
Description: Self-reported number of casual partners in last 3 months among HIV-/u cohort.
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Full Range); unit: Mean of Casual Partners
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 49 | 55 | 57
Mean of Casual Partners | 1.25 [0 to 4] | 1.25 [0 to 4] | 1.33 [0 to 4]

10. Secondary Outcome: HIV Risk Behavior - Reduction in Sexual Partners
Description: Self-reported number of casual partners in last 3 months among HIV-/u cohort.
Time Frame: 12 months
Population: as for outcome 8
Measure: Mean (Full Range); unit: Mean of Casual Partners
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 59 | 72 | 65
Mean of Casual Partners | 1.09 [0 to 4] | 1.15 [0 to 4] | 1.14 [0 to 4]

11. Secondary Outcome: HIV Risk Behavior - Increases in Condom Use
Description: HIV-/u AGYW who reported always using condoms with casual partners in past 3 months.
Time Frame: Baseline
Population: Zambian Adolescent and Young Women not living with HIV. Questions related to sexual behavior and activity can only be asked to individuals aged 15 and over in Zambia. Our HIV-/u cohort is the cohort that enrolled participants between the ages of 10 and 26 and would, therefore, be most affected by the age restrictions in place for sexual behavior questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 14 | 21 | 16
Participants | 3 | 4 | 8

12. Secondary Outcome: HIV Risk Behavior - Increases in Condom Use
Description: HIV-/u AGYW who reported always using condoms with casual partners in past 3 months.
Time Frame: 6 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 8 | 8 | 6
Participants | 7 | 4 | 3

13. Secondary Outcome: HIV Risk Behavior - Increases in Condom Use
Description: HIV-/u AGYW who reported always using condoms with casual partners in past 3 months.
Time Frame: 12 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 11 | 13 | 14
Participants | 2 | 5 | 7

14. Secondary Outcome: HIV Early Detection
Description: HIV-/u proportion with HIV identified through voluntary testing.
Time Frame: 12 months
Population: Zambian Adolescent and Young Women not living with HIV. The 12-month data collection occurred after COVID-19 restrictions had been lifted. The participant count increases from the 6-month count because we were able to contact participants we had previously been unable to reach and participants had moved back to their original enrollment catchment area and could be included in the participant count.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 153 | 147 | 145
Participants | 2 | 2 | 1

15. Secondary Outcome: Linkages to HIV Care - Enrollment at HIV Clinic
Description: Proportion enrolled at an HIV clinic in ≤ 30 days
Time Frame: 6 months
Reporting Status: Not Posted

16. Secondary Outcome: Linkages to HIV Care - Enrollment at HIV Clinic
Description: Proportion enrolled at an HIV clinic in ≤ 30 days
Time Frame: 12 months
Reporting Status: Not Posted

17. Secondary Outcome: Linkages to HIV Care - ART Initiation
Description: Proportion with ART initiated in ≤ 90 days
Time Frame: 6 months
Reporting Status: Not Posted

18. Secondary Outcome: Linkages to HIV Care - ART Initiation
Description: Proportion with ART initiated in ≤ 90 days
Time Frame: 12 months
Reporting Status: Not Posted

19. Secondary Outcome: Adherence to ART
Description: AGYW living with HIV who self-reported "Excellent" medication adherence.
Time Frame: 6 months
Population: Zambian Adolescent and Young Women living with HIV. The 6-month data collection was impacted by the COVID-19 pandemic and restrictions that were in place. We were unable to contact all of the participants we had enrolled at baseline as a result of pandemic restrictions which also caused participants to move away from their original enrollment catchment area. The reduction in participants should not be interpreted as drop-outs or those lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 137 | 138 | 148
Participants | 69 | 83 | 93

20. Secondary Outcome: Adherence to ART
Description: AGYW living with HIV who self-reported "Excellent" medication adherence.
Time Frame: 12 months
Population: Zambian Adolescent and Young Women living with HIV. The 12-month data collection occurred after COVID-19 restrictions had been lifted. The participant count increases from the 6-month count because we were able to contact participants we had previously been unable to reach and participants had moved back to their original enrollment catchment area and could be included in the participant count.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | SHIELD Only | SHIELD + IWC Clinic
Number analyzed (Participants) | 152 | 145 | 145
Participants | 71 | 71 | 84

ADVERSE EVENTS:
Time Frame: 14 months in total
Description: Adverse Events Among Adolescent Girls and Young Women in the SHIELD Study. See note in "Results Participant Flow" and remove all mentions of other phases other than Phase 2 for that is the clinical trial phase. We only have all-cause mortality in this study. The correct all-case mortality numbers can be found below. The reason for the change is that one death involves an individual originally recruited into the HIV-/u cohort and during the course of the intervention became HIV+.
Groups:
- Control HIV+ Caregivers: Caregivers selected by HIV+ AGYW in the control arm.
- SHIELD HIV+ Caregivers: Caregivers selected by HIV+ AGYW in the SHIELD only arm.
- SHIELD HIV- AGYW: HIV- AGYW allocated to the SHIELD only arm.
- SHIELD HIV- Caregivers: Caregivers selected by HIV- AGYW in the SHIELD only arm.
- SHIELD+IWC HIV+ AGYW: HIV+ AGYW allocated to the SHIELD+IWC arm.
- SHIELD+IWC HIV+ Caregivers: Caregivers selected by HIV+ AGYW in the SHIELD+IWC arm.
Arm/Group | Control HIV+ AGYW | Control HIV+ Caregivers | Control HIV- AGYW | Control HIV- Caregivers | SHIELD HIV+ AGYW | SHIELD HIV+ Caregivers | SHIELD HIV- AGYW | SHIELD HIV- Caregivers | SHIELD+IWC HIV+ AGYW | SHIELD+IWC HIV+ Caregivers | SHIELD+IWC HIV- AGYW | SHIELD+IWC HIV- Caregivers
All-Cause Mortality (participants affected / at risk) | 3/177 | 0/154 | 3/198 | 0/194 | 3/171 | 0/150 | 0/201 | 0/197 | 1/175 | 0/139 | 0/201 | 0/193
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/154 | 0/198 | 0/194 | 0/171 | 0/150 | 0/201 | 0/197 | 0/175 | 0/139 | 0/201 | 0/193
Other Adverse Events (participants affected / at risk) | 0/177 | 0/154 | 0/198 | 0/194 | 0/171 | 0/150 | 0/201 | 0/197 | 0/175 | 0/139 | 0/201 | 0/193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03995953/Prot_SAP_000.pdf